CLINICAL TRIAL: NCT03626493
Title: A Research on Hidden Blood Loss in Laparoendoscopic Single-site Radical Hysterectomy With Pelvic Lymphadenectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2018-07-131
Record Dates: First submitted 2018-08-06; First posted 2018-08-13 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Hidden Blood Loss; Single-site Laparoscopy; Radical Hysterectomy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LSRH: patients who undergo laparoendoscopic single-site radical hysterectomy with pelvic lymphadenectomy

SUMMARY:
The aim of this cross-sectional study is to evaluate the hidden blood loss in patients who undergo laparoendoscopic single-site radical hysterectomy with pelvic lymphadenectomy and identity its risk factors.

DETAILED DESCRIPTION:
The electronic medical data of 105 patients who undergo laparoendoscopic single-site radical hysterectomy in the following year to treat cervical cancer will be analyzed retrospectively in this study. The amount of hidden blood loss will be calculated according to Gross's formula. And multiple linear regression analysis will be employed to identify its risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the study with informed consent;
2. Females aged 20-80 who are confirmed with cervical cancer and are treated with laparoendoscopic single-site radical hysterectomy with pelvic lymphadenectomy.

Exclusion Criteria:

1. Pregnancy, lactation, postmenopause, or planned pregnancy within two years;
2. Suspected or identified as other tumors of genital tract;
3. History of hyperparathyroidism, infectious diseases (tuberculosis, AIDS), autoimmune diseases, or digestive system diseases (malabsorption, crohn disease and dysentery);
4. Other diseases or heavy injuries that will interfere with the results;
5. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The planned sample size was based on data from a previous study, in which the standard deviation was 5. We assumed an one-tailed α error of 0.05 and a sampling error of 1.0. we propose to enroll 105 participants and allow for a dropout rate of 10% for an effective sample size of 100.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
the volume of hidden blood loss (mL) | 10 months after the operation
  the specific volume of hidden blood loss in patients after the operation applying Gross's formula

SECONDARY OUTCOMES:
the risk factors of hidden blood loss | 10 months after the operation
  Performing multiple linear regression analysis with SPSS 17.0, we plan to identify the risk factors which can increase the volume of hidden blood loss from possible factors like hypertension, diabetes, etc.
the volume of total blood loss (mL) | 10 months after surgery
  the volume of blood loss happened to patients through the whole perioperative period accoring to the method of Nadler
the volume of visible blood loss (mL) | 10 months after surgery
  the volume of visible blood loss including the blood in the suction bottle and in weighed compresses during the operation and the drainage volume as the post-operative blood loss

CONTACTS AND LOCATIONS:
Locations (1):
- TING LI, Wenzhou, Zhejiang, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03626493/Prot_SAP_000.pdf